CLINICAL TRIAL: NCT00348790
Title: A Phase II Trial of PTK-787 in Recurrent or Progressive Meningiomas
Brief Title: Vatalanib in Treating Patients With Recurrent or Progressive Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jeffrey Raizer, Jeffrey Raizer, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05C4; STU00005338 (Other: Northwestern University IRB); NU 05C4 (Other: Northwestern University)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Brain and Central Nervous System Tumors; Sarcoma
Keywords: adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult malignant hemangiopericytoma; adult anaplastic meningioma; adult papillary meningioma; adult melanocytic lesion; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Sarcoma; Meningioma; Hemangiopericytoma, Malignant; Brain Neoplasms | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vatalanib (Experimental): Patients will be treated with 500 mg of vatalanib, administered orally, twice a day for 28 days (1 cycle). Patients will start at a dose of 250 mg twice a day and increase by 250 mg per day every 7 days until 500 mg twice a day is reached.
  Patients who are responding may remain on study treatment for 12 months.
  Interventions: Drug: vatalanib

INTERVENTIONS:
Drug: vatalanib
  Other Names: PTK787; ZK 222584

SUMMARY:
RATIONALE: Vatalanib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well vatalanib works in treating patients with recurrent or progressive meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of vatalanib, in terms of radiographic improvement and clinical improvement, in patients with recurrent or progressive meningioma.

Secondary

* Determine the 6-month progression-free survival of these patients.
* Describe the response rate and overall survival of these patients.
* Determine the safety of vatalanib in these patients.
* Correlate the response rates with expression of vascular endothelial growth factor, epidermal growth factor receptor, platelet-derived growth factor, and HER2.
* Develop exploratory data concerning surrogate markers of angiogenic activity in vivo using magnetic resonance perfusion.

OUTLINE: Patients receive oral vatalanib twice daily on days 1-28. Courses repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 1 year.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed meningioma, including the following subtypes:

  * Benign meningioma
  * Malignant meningioma

    * Steroid dosage stable for ≥ 5 days
  * Atypical meningiomas
  * Hemangiopericytoma
* May or may not have neurofibromatosis (NF) type 1 or 2 disease

  * Patients with a history of NF may have other stable CNS tumors, such as schwannoma, acoustic neuroma, or ependymoma only if those lesions have been stable for the past 6 months
* Progressive or recurrent disease by MRI or CT scan

  * Prior radiotherapy allowed provided evidence of disease progression is documented by positron emission tomography, thallium scanning, magnetic resonance spectroscopy, or surgery to rule out radiation necrosis for patients treated with radiosurgery
* Recent resection of recurrent or progressive tumor allowed provided both of the following criteria are met:

  * At least 4 weeks since prior surgery and recovered
  * Evaluable residual disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* SGOT and SGPT < 2 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine < 1.5 mg/dL
* Negative proteinuria dipstick OR total urinary protein ≤ 500 mg AND creatinine clearance ≥ 50 mL/min
* PT, INR, and PTT ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 6 months after completion of study treatment
* No history of any other cancer except nonmelanoma skin cancer or carcinoma in situ of the cervix, unless in complete remission and off all therapy for that disease for ≥ 3 years
* No disease that would obscure toxicity or dangerously alter drug metabolism
* No bleeding disorders
* No severe and/or uncontrolled medical conditions that would limit compliance with study requirements, including any of the following:

  * Uncontrolled high blood pressure
  * History of labile hypertension
  * History of poor compliance with an antihypertensive regimen
  * Unstable angina pectoris
  * Symptomatic congestive heart failure
  * Myocardial infarction within the past 6 months
  * Serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes
  * Active or uncontrolled infection
  * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
  * Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of vatalanib (i.e., ulcerative disease, uncontrolled nausea, vomiting, or diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow tablets)
  * QTc > 450 (male) or > 470 (female)
  * Congenital or acquired long QTc syndrome

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 4 weeks since prior radiotherapy, including external-beam radiotherapy, interstitial brachytherapy, or gamma-knife radiosurgery
* At least 4 weeks since prior investigational agents
* More than 4 weeks since prior cytotoxic therapy (6 weeks for nitrosoureas)
* More than 4 weeks since prior immunotherapy
* More than 2 weeks since prior noncytotoxic or biologic therapies
* At least 2 weeks since prior drugs that affect hepatic metabolism (steroids should be tapered off if not clinically indicated)
* At least 2 weeks since prior and no concurrent enzyme-inducing anticonvulsant drugs
* No prior antivascular endothelial growth factor therapy
* No other concurrent investigational agents or anticancer therapy (including chemotherapy, radiotherapy, hormonal therapy, or immunotherapy)
* No concurrent warfarin
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-05; Primary Completion 2010-11 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Began Treatment
Arm/Group | Vatalanib
Started | 25
Completed | 25
Not Completed | 0
Period: Completed Treatment
Arm/Group | Vatalanib
Started | 25
Completed | 0
Not Completed | 25
Not completed — Withdrawal by Subject | 4
Not completed — Disease progression | 14
Not completed — Adverse Event | 4
Not completed — Required surgery | 2
Not completed — Unable to travel to study site | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vatalanib
Number analyzed (Participants) | 25
Age, Customized [Number; unit: participants]
  21-30 | 1
  31-40 | 1
  41-50 | 6
  51-60 | 8
  61-70 years | 8
  71-80 | 0
  81-90 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who DID NOT Experience Disease Progression or Death by 6 Months After Starting Treatment.
Description: Patients were assessed with imaging techniques (MRI) during screening/baseline and then every 2 months after starting treatment. Survival status and disease status were recorded. The number of patients who did not experience an event (defined as either death for any reason or progression of their disease) by 6 months after starting treatment were counted.
Time Frame: From the date the first patient began treatment until the date the last patient has disease progression, becomes deceased, or completes 6 months of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vatalanib
Number analyzed (Participants) | 25
Participants | 15

2. Secondary Outcome: Determine Efficacy (Radiographic and Clinical Improvement)
Description: Efficacy will be assessed by MRI scan and neurological exam upon study entry, every 2 weeks for 2 months, then every 8 weeks while on treatment
Time Frame: At baseline, every 2 weeks for 2 months, then every 8 weeks while on treatment
Population: Data not collected. Statistical design of study was based on participation of patients with WHO grade I meningioma. Most patients enrolled in the study were WHO grade II and WHO grade III.
Groups:
- Vatalanib: Patients will be treated with 500 mg of vatalanib, administered orally, twice a day for 28 days (1 cycle). Patients will start at a dose of 250 mg twice a day and increase by 250 mg per day every 7 days until 500 mg twice a day is reached.
  Patients who are responding may remain on study treatment for 12 months.
  vatalanib
Arm/Group | Vatalanib
Number analyzed (Participants) | 0

3. Secondary Outcome: Best Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) will be as assessed by MRI scan every 2 months while on study treatment and follow-up for up to 1 year after discontinuation of study treatment. The RR is the best response recorded from the start of the treatment until disease progression (PD) where the following definitions apply.
  Complete Response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions.
  Partial Response (PR): Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
  Stable/No Response: Does not qualify for CR, PR, or PD Progressive disease (PD):25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) worsening of evaluable disease, new lesions, clinical worsening OR failure to return for evaluation due to death/deteriorating condition
Time Frame: Every 2 months for up to 1 year after study treatment.
Population: 3 patients not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Vatalanib
Number analyzed (Participants) | 22
Participants
  SD | 15
  SD on MRI but clinical decline | 2
  PD | 5

4. Secondary Outcome: To Correlate the Response Rates With Expression of Certain Types of Genes
Description: Correlation of response rates with the expression of certain types of genes will be assessed by examining tissue samples taken from previous surgery and testing for certain genes
Time Frame: At the end of study treatment
Population: Data not collected and analyzed.
Arm/Group | Vatalanib
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety of Vatalanib in Patients With Recurrent of Progressive Meningiomas
Description: Safety of vatalanib will be assessed using National Cancer Institute Common Terminology Criteria of Adverse Events (NCI CTCAE) 3.0 and graded using the following:
  Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Fatal
Time Frame: Every week while on study treatment until 30 days after last treatment.
Population: Toxicities determined to be either grade 3 or grade 4 and at least possibly related to study drug are reported here.
Measure: Number; unit: participants
Arm/Group | Vatalanib
Number analyzed (Participants) | 25
participants
  Dehydration | 1
  Deep vein thrombosis | 1
  Fatigue | 4
  Gastrointestinal | 1
  Hypertension | 1
  Hyponatremia | 1
  Leukopenia | 1
  Pain | 1
  Rash | 1
  Transaminase | 2
  Weight loss | 1

6. Secondary Outcome: Number of Months Patients Survive After Being Treatment on the Study.
Time Frame: From the date the first patient began treatment until the date the last patient became deceased.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vatalanib
Number analyzed (Participants) | 25
months | 29.2 [15 to 50]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival will be measured from the first treatment on study until death of any cause.
Time Frame: Every 2 months for up to 1 year after study treatment.
Population: Number of patients with WHO grade II or WHO grade III meningioma.
Measure: Median (Full Range); unit: Months
Arm/Group | Vatalanib
Number analyzed (Participants) | 21
Months | 26 [4.27 to 76.75]

8. Other Pre Specified Outcome: Develop Data Concerning Certain Genes That Cause Tumors to Grow New Blood Vessels
Description: Data concerning certain genes that cause tumors to grow new blood vessels will be examined by MRI scan with MR Perfusion done before treatment and then every 2 months while on study treatment
Time Frame: MRI with MR Perfusion will be done before treatment and then every 2 months while on study treatment
Population: Data not collected and analyzed.
Arm/Group | Vatalanib
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: To Use the FACT BR Questionnaire to Measure Quality of Life
Description: FACT BR questionnaire will be used to measure quality of life at baseline and then every time an MRI scan is performed while on study treatment
Time Frame: At baseline and then every time an MRI is performed while on study treatment.
Population: Data not collected or analyzed.
Arm/Group | Vatalanib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Patients were assessed for adverse events every 2 weeks for the first 2 months, then every 4 weeks (monthly) while on treatment and up to 30 days after the final dose of study drug.
Arm/Group | Vatalanib
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vatalanib (N=25)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1 — Subject was admitted for elective craniotomy. Subject went into atrial fibrillation unrelated to study drug.
Rash (Skin and subcutaneous tissue disorders) | 1
Scalp wound (Skin and subcutaneous tissue disorders) | 1 — Subject was admitted after falling with scalp wound. The injury was unrelated to study treatment.
Vertigo (Ear and labyrinth disorders) | 1
Nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vatalanib (N=25)
Anemia (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 5
Hypertension (Cardiac disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 3
Fatigue (General disorders) | 19
Neuropathy: Sensory-facial (Nervous system disorders) | 4
Neuropathy - Motor (Nervous system disorders) | 4
Pain (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 12
Weight loss (Investigations) | 3
Transaminase (Metabolism and nutrition disorders) | 15
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 2
Insomnia (General disorders) | 5
T wave abnormalities/changes (Cardiac disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2
Depression (Psychiatric disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Seizure (Nervous system disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Vision loss (Eye disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Proteinuria (Metabolism and nutrition disorders) | 5
Sinus tachycardia (Cardiac disorders) | 2
Memory impairment (Nervous system disorders) | 2
Spasm (Nervous system disorders) | 3
Confusion (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes